CLINICAL TRIAL: NCT02607163
Title: The Effect of Dexmedetomidine on Prevention of Postoperative Acute Kidney Injury in Patients Undergoing Aortic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 4-2015-0672
Record Dates: First submitted 2015-11-15; First posted 2015-11-17 (Estimated); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Acute Kidney Injury(Postoperative Acute Kidney Injury in Patients Undergoing Aortic Surgery)
MeSH Terms: interventions — Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- dexmedetomidine (Experimental): dexmedetomidine, 0.4 mcg/kg/h, IV, The infusion of study drug is started after anesthesia induction and continued until 24 hours after surgery.
  Interventions: Drug: dexmedetomidine
- control (Placebo Comparator): saline, same infusion rate (received equal volume of normal saline), IV, The infusion of study drug is started after anesthesia induction and continued until 24 hours after surgery.
  Interventions: Drug: saline

INTERVENTIONS:
Drug: dexmedetomidine — Immediately after the induction of anesthesia, patients in the dexmedetomidine group received dexmedetomidine continuous intravenous (IV) infusion of 0.4 mcg/kg/h until 24 hours after surgery.
  Arms: dexmedetomidine
Drug: saline — same infusion rate (received equal volume of normal saline), IV, The infusion of study drug is started after anesthesia induction and continued until 24 hours after surgery.
  Arms: control

SUMMARY:
Acute kidney injury(AKI) is a common and severe complication after the cardiac surgery. Postoperative AKI increases the in-hospital stay, intensive care unit(ICU) stay and postoperative mortality. Aortic surgery is the most risky surgery that causes the postoperative AKI, and the incidence of AKI after aortic surgery is about 50%.

The α1- and α2-adrenergic receptors in the kidney modulate vasoconstrictor and vasodilatory effects, respectively. Agents that attenuate renal vasoconstriction may have potential as renoprotective drugs because vasoconstriction most likely contributes to the pathophysiology of AKI. Clonidine, an α2-agonist, has been shown experimentally to inhibit renin release and cause a diuresis, and it has been evaluated in an experimental AKI model, confirming its potential as a renoprotective agent. Furthermore, it has been already reported that dexmedetomidine, α2-agonist, reduce the impairment of renal function after cardiac operation.

The aim of this study is to examine the association between preoperative dexmedetomidine infusion and the incidence of postoperative acute kidney injury(AKI) in patients undergoing aortic surgery.

ELIGIBILITY:
Inclusion Criteria:

1. the patients undergoing ascending, arch and/or proximal descending aorta surgery with cardiopulmonary bypass
2. 20 - 100 yrs old

Exclusion Criteria:

1. having preoperative severe renal dysfunction (eGFR < 15 ml/min per 1.73m2)
2. Left ventricular-ejection fraction < 30%
3. Preexisting congestive heart failure
4. Severe coronary artery disease
5. Hemodynamically unstable arrhythmia
6. Cardiogenic shock during perioperative period
7. Ventricular assist device use
8. cannot communication because of a language barrier or illiteracy

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2019-03-06 (Actual); Study Completion 2019-03-06 (Actual)

PRIMARY OUTCOMES:
Acute kidney injury (AKI) after aortic surgery (AKI according to the Kidney Disease Improving Global Outcomes (KDIGO) criteria) | up to 7 days after the aortic surgery
  0.3 mg/dl increase in serum creatinine concentration within 48 hours OR, a 50% increase within 7 days postoperatively OR, urine volume < 0.5 ml/kg/h for 6 hours

SECONDARY OUTCOMES:
Acute kidney injury (AKI) after aortic surgery (AKI according to the Kidney Disease Improving Global Outcomes (KDIGO) criteria) | up to 7 days after the surgery
  KDIGO stage 2: Serum creatinine increase to 2-3-fold from baseline OR urine output < 0.5 ml/kg/h for 12h
Acute kidney injury (AKI) after aortic surgery (AKI according to the Kidney Disease Improving Global Outcomes (KDIGO) criteria) | up to 7 days after the surgery
  KDIGO stage 3: Serum creatinine increase to 3.0-fold from baseline OR Increase in serum creatinine to ≥ 4 mg/dl OR Initiation of renal replacement therapy OR In patients <18 years, decrease in eGFR to < 35 ml/min per 1.73 m2 OR Anuria for ≥ 12h.
major morbidity endpoint | acute kidney injury - up to 7 days after the surgery; Other - during the hospitalization for surgery
  acute kidney injury (same as the primary endpoint), permanent stroke, prolonged ventilator care >24h, deep wound infection, and mortality.
postoperative delirium | up to 7 days after the surgery
  delirium - assessed with The American Psychiatric Association's fifth edition of the Diagnostic and Statistical Manual of Mental Disorders or Confusion Assessment Method for the ICU
drug-related adverse events | hypotension or bradycardia: during surgery; Other - during surgery and 24 hours after surgery
  hypotension (mean arterial pressure <60 mmHg) or bradycardia (<50 beats/min) OR the use of vasopressor, inotropes or temporary pacing, OR postoperative arrhythmia

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yonsei Cardiovascular Hospital, Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Derived] Soh S, Shim JK, Song JW, Bae JC, Kwak YL. Effect of dexmedetomidine on acute kidney injury after aortic surgery: a single-centre, placebo-controlled, randomised controlled trial. Br J Anaesth. 2020 Apr;124(4):386-394. doi: 10.1016/j.bja.2019.12.036. Epub 2020 Jan 29. PMID 32007239